CLINICAL TRIAL: NCT01666379
Title: Pain Management After Forefoot Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Riika Merivirta, M.D., Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ForefootFenta vs.2
Record Dates: First submitted 2012-07-19; First posted 2012-08-16 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Postoperative Pain
Keywords: Hallux valgus; Forefoot; transdermal fentanyl
MeSH Terms: conditions — Pain, Postoperative; Hallux Valgus | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fentanyl (Experimental)
  Interventions: Drug: Fentanyl
- placebo (Placebo Comparator)

INTERVENTIONS:
Drug: Fentanyl
  Arms: Fentanyl

SUMMARY:
The purpose of this study was to compare the efficacy of transdermal fentanyl to placebo both administered together with peroral nonsteroidal antiinflammatory drug (NSAID) and paracetamol in treatment of postoperative pain after hallux valgus or hallux rigidus surgery.

ELIGIBILITY:
Inclusion Criteria:

* unilateral hallux valgus or hallux rigidus surgery
* 18-75 yrs old
* ASA I-III

Exclusion Criteria:

* previous history of intolerance to the study drug
* history of alcoholism
* drug abuse
* psychological or other emotional problems that are likely to invalidate informed consent
* sleep apnoea
* BMI ≥ 35 kg/m2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Consumption of rescue opioid | on the 1st postoperative day
  Also adverse effects were evaluated but this evaluation was not the first or secondary outcome measure

SECONDARY OUTCOMES:
Pain on a numerical scale | on the 1st postoperative day
  The adverse effects were evaluated but the evaluation was not the first or secondary outcome measure

CONTACTS AND LOCATIONS:
Locations (1):
- The Department of Anaesthesiology, Intensive Care, Emergency Care and Pain Management of Turku University Hospital, Turku, Finland